CLINICAL TRIAL: NCT02736916
Title: Hippocampal-Sparing Whole-Brain Radiation Therapy for Prophylactic Cranial Irradiation in Limited Stage Small Cell Lung Cancer
Brief Title: HS-WBRT for Prophylactic Cranial Irradiation in Limited Stage Small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Radiation Oncology 20160101
Record Dates: First submitted 2016-03-25; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Small Cell Lung
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HS-WBRT PCI (Experimental): LD-SCLC patients with HS-WBRT PCI
  Interventions: Radiation: HS-WBRT PCI
- Conventional PCI (Active Comparator): LD-SCLC patients with Conventional PCI
  Interventions: Radiation: Conventional PCI

INTERVENTIONS:
Radiation: HS-WBRT PCI — LD-SCLC patients with HS-WBRT PCI
  Arms: HS-WBRT PCI
Radiation: Conventional PCI — LD-SCLC patients with conventional PCI
  Arms: Conventional PCI

SUMMARY:
Prophylactic cranial irradiation (PCI) is an important treatment modality of patients with limited stage small cell lung cancer (LD-SCLC). However, PCI is also associated with several side effects, such as decline in memory and other cognitive functions. This provides the rationale to explore the clinical feasibility of hippocampal avoidance during WBRT. Previous studies have demonstrated the dosimetric capabilities of IMRT to conformally avoid the hippocampus without detriment to the radiation dose the remaining brain receives. The aims of this study is to evaluate the therapy efficacy and the safety profile of hippocampal-sparing whole-brain radiation therapy (HS-WBRT) for PCI in patients with LD-SCLC.

DETAILED DESCRIPTION:
Chemotherapy plus thoracic radiation followed by prophylactic cranial irradiation (PCI) is the standard of care in management of limited stage small cell lung cancer patients. However, whole brain radiation therapy (WBRT) is also associated with many side effects including consolidation of new memory, poor attention span/concentration, visual spatial difficulties, difficulty with executive planning, and poor fine motor control. There exists significant preclinical and clinical evidence that radiation induced injury to the hippocampus correlates with neurocognitive decline of patients who received WBRT. Reducing radiation dose to the hippocampus during WBRT has been postulated as an approach to mitigate neurocognitive impairment. The present study hypothesize that hippocampal sparing PCI will allow improved performance on tests of short term memory and executive function compared to a historical control receiving the same dose of conventional PCI. The primary objective of this study is to evaluate performance on the Hopkins Verbal Learning Test-Revised for delayed recall at 6 months following hippocampal-sparing PCI relative to the historical control. Secondary objectives are to estimate: composite cognitive function following hippocampal-sparing PCI relative to the historical control and the rate of metastases in the hippocampus at 2 years following hippocampal-sparing PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have newly diagnosed and confirmed small-cell lung cancer (SCLC)
* Patient must have a performance status of 1 or higher
* Patients must not have received previous irradiation to the brain
* Patients must have limited stage disease with CR (complete response) to chemotherapy and consolidative chest radiotherapy that was documented at least on standard chest x-rays within one month of study entry
* Negative MRI or CT scan of the brain at least one month before protocol entry
* Women of child-bearing potential must have a negative pregnancy test and also agree to use adequate contraceptives while on protocol
* Patient must be able to understand and sign the informed consent document
* Patient must be informed of the investigational aspect to this trial prior to singing the informed consent document

Exclusion Criteria:

* Patients receiving prior external beam irradiation to the head or neck, including any form of stereotactic irradiation
* Radiographic evidence of brain metastases and/or ipsilateral lung metastases/malignant pleural effusion
* Planned concurrent chemotherapy or antitumoral agent during PCI
* Concomitant malignancy or malignancy within the past five years other than nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Patients with minimal pleural effusion evident on CXR (chest X-ray); minimal pleural effusion visible on chest CT is allowed.
* Patients with epilepsy requiring permanent oral medication _ Patients must not have a serious medical or psychiatric illness that would, in the opinion of the investigator, prevent informed consent or completion of protocol treatment, and/or follow-up visits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate delayed recall as assessed by the Hopkins Verbal Learning Test-Revised (HVTL-R) 4 months after hippocampal sparing during whole-brain radiotherapy (HS-WBRT) for PCI of limited stage small cell lung cancer patients. | The change of the performance on the Hopkins Verbal Learning Test-Revised for delayed recall at 4 months following hippocampal-sparing PCI relative to the control group

SECONDARY OUTCOMES:
Evaluate the rate of brain metastasis in hippocampal region after HS-WBRT PCI for limited stage small cell lung cancer patients. | The metastatic rate between HS-WBRT and control group at 2 years following hippocampal-sparing PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Zhao, M.D., Study Chair — General Hospital of Ningxia Medical Universuty
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No